CLINICAL TRIAL: NCT07140822
Title: A Prospective, Multi-center, Non-inferiority and Randomized Controlled Clinical Study to Evaluate the Safety and Effectiveness of the Coronary Cutting Balloon Catheter in the Treatment of Coronary Artery Disease (CAD)
Brief Title: A Randomized Study of Cutting Balloon Catheter for CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCBP01
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention (PCI); Calcified Coronary Lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary Cutting Balloon Catheter (Experimental)
  Interventions: Device: Coronary Cutting Balloon Catheter
- VesscideTM Cutting Balloon System (Active Comparator)
  Interventions: Device: VesscideTM Cutting Balloon System

INTERVENTIONS:
Device: Coronary Cutting Balloon Catheter — This product uses a pressure device to pressurize the balloon to expand it. The blades designed on the surface of the balloon produce a cutting effect on the vascular lesions, allowing it to better embed into the plaque.
  Arms: Coronary Cutting Balloon Catheter
Device: VesscideTM Cutting Balloon System — This product utilizes a pressure mechanism to inflate the balloon, causing it to expand. The blades on the balloon's surface create a cutting action on the vascular lesions, enabling the device to penetrate the plaque more effectively.
  Arms: VesscideTM Cutting Balloon System

SUMMARY:
This study is designed as a prospective, multi-center, non-inferiority and randomized controlled clinical trial. A total of 158 eligible subjects from 18 sites across the country is planned to be enrolled, and they will be randomly assigned to the test group and the control group according to a ratio of 1:1 for balloon dilatation for the treatment of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-80 years, including 18 and 80 years;
* Patients with stable or unstable angina, or old myocardial infarction or clinically judged silent myocardial ischemia (target vessel reference vessel diameter 2.00-4.00 mm (both inclusive)), luminal diameter stenosis ≥ 70%, or ≥ 50% by visual inspection with evidence of ischemia, TIMI blood flow ≥ grade 1, and requiring treatment with a cutting balloon dilatation catheter as considered by the operator;
* Able to understand the purpose of the study, participate the study willingly, sign the written informed consent form, and are available for and willing to follow-up as defined in this trial.

General exclusion criteria:

1. Pregnant or lactating women or women who are planning pregnancy;
2. Subjects with myocardial infarction occurred within one week; the myocardial enzyme TNI or TNT has not returned to normal although myocardial infarction has occurred for more than one week;
3. Subjects who are considered by the investigator through angiography that the cutting balloon cannot pass through even dilatation with a small one and need a rotational atherectomy;
4. Non-target vessels, which can be treated simultaneously with the target blood vessel, have not been treated well in advance, or the total number of lesions on the non-target blood vessel is > 3;
5. NYHA Class IV patients;
6. Patients with severe renal failure (creatinine > 443 μmol/L) or ongoing hemodialysis therapy;
7. Heart transplant patients;
8. Patients with graft vessel disease;
9. Patients with hemodynamic instability or symptoms of shock;
10. Patients with a life expectancy of no more than 1 year;
11. Patients who are expected to undergo elective surgery within 1 month;
12. Patients not eligible for coronary artery bypass grafting (CABG) procedure;
13. Patients with a predisposition to bleeding, a history of active peptic ulcer, or contraindications to antiplatelet agents and anticoagulants, patients who cannot undergo anticoagulant therapy, or patients who have experienced hemorrhagic stroke within 6 months;
14. Patients who are known to be allergic or contraindicated to heparin, contrast agents, etc.;
15. Patients who are suffering from diseases that can cause difficulties in treatment and evaluation;
16. Patients who have been selected and have participated in trials with other drug or medical device but have not reached the time limit of the primary study endpoint;
17. Clinicians expect that the risk of interventional surgery is extremely high or other cases that should be ruled out;
18. Patients who, in the judgment of the investigator, are poor compliance with the therapy and are unable to complete the trial as required;

    Lesion related exclusion criteria:
19. Left main lesion or lesion at a distance of ≤ 2 mm from the left main coronary artery;
20. Patients with thrombosis suggested by angiography;
21. Patients with a total occluded lesion and a TIMI flow grade 0;
22. Coronary artery spasm (CAS) without organic stenosis;
23. Left main lesion without protection from bypass grafts or collateral flow;
24. In addition to the above contraindications, conditions diagnosed by the physician as unsuitable for the use of the device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Acute gain | Before and after balloon dilation
  The acute gain is defined as the difference in minimal lumen diameter (MLD) of the target lesions measured by quantitative coronary angiography (QCA) before and after the balloon dilatation using balloons from the test group/control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Meizhou People's Hospital, Meizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No